CLINICAL TRIAL: NCT03730649
Title: Effect of Topical Sulforaphane on Skin Aging and With Ultraviolet and Visible Light Exposure
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00184806
Record Dates: First submitted 2018-11-02; First posted 2018-11-05 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Skin Aging
MeSH Terms: interventions — sulforaphane; Light

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sulforaphane without light challenge (Active Comparator): Participants with moderate photodamage and moderate intrinsic skin aging will apply sulforaphane (broccoli sprout extract) in jojoba oil nightly (without any UV or visible light irradiation) for up to 6 months and have up to 9 biopsies taken just before treatment and occurring at regular intervals during the study
  Interventions: Drug: Sulforaphane (broccoli sprout extract)
- Sulforaphane with light challenge (Active Comparator): Participants will have 2 test areas irradiated with up to 5 UV or visible light treatments and biopsies taken before and within 7 days after UV or visible light irradiation; one of the UV/visible light treated areas will be pre-treated with sulforaphane (broccoli sprout extract) for up to 28 consecutive nights and the other UV/visible light treated areas will be pre-treated with jojoba oil.
  Interventions: Drug: Sulforaphane (broccoli sprout extract); Radiation: UV or visible light

INTERVENTIONS:
Drug: Sulforaphane (broccoli sprout extract) — Participants will topically apply Sulforaphane for a period of time
Radiation: UV or visible light — Participants will have 2 test areas irradiated with up to 5 UV or visible light treatments
  Arms: Sulforaphane with light challenge

SUMMARY:
The study is to compare the expression of both keratin 16 and 17 before and after application of sulforaphane on both photoprotected and photoexposed area, and to determine whether these findings alter skin aging as well as skin response to ultraviolet (UV) and visible light exposure.

DETAILED DESCRIPTION:
The study is to compare the expression of both keratin 16 and 17 before and after application of sulforaphane on both photoprotected and photoexposed area, and to determine whether these findings alter skin aging as well as skin response to ultraviolet (UV) and visible light exposure.

Each study participant will have up to eight study visits. Topical sulforaphane will be applied for up to 6 months. Photography, clinical assessment, UV light irradiation, Visible light treatment, Skin biopsies, non invasive elasticity measurements such as cutometer and ballistometer, and others will be involved in this study.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be over the age of 18 years old with healthy skin or moderate degree of photoaging/intrinsic aging;
* Must be healthy enough to undergo skin biopsy, light irradiation, and other study procedures in the opinion of the investigator;
* Must be willing to comply with the requirements of the protocol;
* Must have the ability to understand and communicate with the investigator;
* Participant must provide informed consent.

Exclusion Criteria:

* Subjects who are unable to provide informed consent;
* Subject with significant medical history or current skin diseases that the investigator feels is not safe for study participation;
* Subjects who have been treated with systemic retinoids or steroids within the past month prior to entry to the study;
* Subjects who have been treated with topical steroids, retinoids or other topical drugs used within 2 weeks prior to entry to the study;
* Recently treated or current skin diseases that would affect clinical evaluation and biopsy;
* Subjects with a known allergy to broccoli.
* Presence or suspicion of bleeding disorder or diathesis which would complicate biopsy.
* Subjects with a history of excessive scar or keloid formation in the past 10 years.
* Pregnant or nursing subjects (self-reported).
* Subjects with known allergy to anesthetics used.
* Patients with history of investigational drug use in the 30 days prior to entry into the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-10-09 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
keratin 16 presence as determined by immunofluorescence assay | Up to 6 months
  The investigators will detect the presence of keratin 16 in the basal layer of the epidermis in both photoprotected and photodamaged skin treated with sulforaphane (SF), by immunofluorescence assay, to determine whether SF can improve skin fragility and other features seen in these conditions
keratin 17 presence as determined by immunofluorescence assay | Up to 6 months
  The investigators will detect the presence of keratin 17 in the basal layer of the epidermis in both photoprotected and photodamaged skin treated with SF, by immunofluorescence assay, to determine whether SF can improve skin fragility and other features seen in these conditions
keratin 16 fold change as determined by Reverse Transcription Polymerase Chain Reaction (RT-PCR) | Up to 6 months
  The investigators will detect the fold change of keratin 16 in the basal layer of the epidermis in both photoprotected and photodamaged skin treated with SF, by RT-PCR, to determine whether SF can improve skin fragility and other features seen in these conditions
keratin 17 fold change as determined by RT-PCR | Up to 6 months
  The investigators will detect the fold change of keratin 17 in the basal layer of the epidermis in both photoprotected and photodamaged skin treated with sulforaphane (SF), by RT-PCR, to determine whether SF can improve skin fragility and other features seen in these conditions

SECONDARY OUTCOMES:
keratin expression changes as determined by RT-PCR | Up to 6 months
  The investigators will test the fold change of keratin expression in human skin after acute UV and visible light light exposure, separately and in combination with application of topical sulforaphane by RT-PCR.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Chien, Principal Investigator — Department of Dermatology, Johns Hopkins School of Medicine
Locations (1):
- Cutaneous Translational Research Program, Department of Dermatology, Johns Hopkins University School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dinkova-Kostova AT, Talalay P, Sharkey J, Zhang Y, Holtzclaw WD, Wang XJ, David E, Schiavoni KH, Finlayson S, Mierke DF, Honda T. An exceptionally potent inducer of cytoprotective enzymes: elucidation of the structural features that determine inducer potency and reactivity with Keap1. J Biol Chem. 2010 Oct 29;285(44):33747-55. doi: 10.1074/jbc.M110.163485. Epub 2010 Aug 26. PMID 20801881
- [Background] Talalay P, Fahey JW, Healy ZR, Wehage SL, Benedict AL, Min C, Dinkova-Kostova AT. Sulforaphane mobilizes cellular defenses that protect skin against damage by UV radiation. Proc Natl Acad Sci U S A. 2007 Oct 30;104(44):17500-5. doi: 10.1073/pnas.0708710104. Epub 2007 Oct 23. PMID 17956979
- [Background] Shapiro TA, Fahey JW, Dinkova-Kostova AT, Holtzclaw WD, Stephenson KK, Wade KL, Ye L, Talalay P. Safety, tolerance, and metabolism of broccoli sprout glucosinolates and isothiocyanates: a clinical phase I study. Nutr Cancer. 2006;55(1):53-62. doi: 10.1207/s15327914nc5501_7. PMID 16965241
- [Background] Egner PA, Chen JG, Wang JB, Wu Y, Sun Y, Lu JH, Zhu J, Zhang YH, Chen YS, Friesen MD, Jacobson LP, Munoz A, Ng D, Qian GS, Zhu YR, Chen TY, Botting NP, Zhang Q, Fahey JW, Talalay P, Groopman JD, Kensler TW. Bioavailability of Sulforaphane from two broccoli sprout beverages: results of a short-term, cross-over clinical trial in Qidong, China. Cancer Prev Res (Phila). 2011 Mar;4(3):384-95. doi: 10.1158/1940-6207.CAPR-10-0296. PMID 21372038
- [Background] Singh K, Connors SL, Macklin EA, Smith KD, Fahey JW, Talalay P, Zimmerman AW. Sulforaphane treatment of autism spectrum disorder (ASD). Proc Natl Acad Sci U S A. 2014 Oct 28;111(43):15550-5. doi: 10.1073/pnas.1416940111. Epub 2014 Oct 13. PMID 25313065
- [Background] Kerns ML, DePianto D, Dinkova-Kostova AT, Talalay P, Coulombe PA. Reprogramming of keratin biosynthesis by sulforaphane restores skin integrity in epidermolysis bullosa simplex. Proc Natl Acad Sci U S A. 2007 Sep 4;104(36):14460-5. doi: 10.1073/pnas.0706486104. Epub 2007 Aug 27. PMID 17724334
- [Background] Sikdar S, Papadopoulou M, Dubois J. What do we know about sulforaphane protection against photoaging? J Cosmet Dermatol. 2016 Mar;15(1):72-7. doi: 10.1111/jocd.12176. Epub 2016 Jan 22. PMID 26799467